CLINICAL TRIAL: NCT05245721
Title: Effect of Caudal Nalbuphine on Postoperative Emergence Agitation in Pediatrics Undergoing Infra-umbilical Surgeries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Adel Ebrahim Okely, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17101501
Record Dates: First submitted 2022-01-18; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Agitation, Emergence; Post Operative Pain
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative | interventions — Nalbuphine; Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nalbuphine (Active Comparator)
  Interventions: Drug: Nalbuphine; Drug: Bupivacain
- Bupivacaine (Active Comparator)
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Nalbuphine — Caudal nalbuphine injection in pediatrics undergoing infra-umbilical surgeries
  Arms: Nalbuphine
Drug: Bupivacain — Caudal bupivacaine in pediatrics undergoing infra-umbilical surgeries

SUMMARY:
Effect of caudal nalbuphine on postoperative emergence agitation in pediatrics undergoing infra-umbilical surgeries and pain assessment

ELIGIBILITY:
Inclusion Criteria:

* Age 2_12 years
* Both genders
* ASA I_II
* Children undergoing infra-umbilical surgeries

Exclusion Criteria:

* Guardians refusal
* congenital anomalies at the lower spine or meringues
* Increased intracranial pressure
* Skin infection at site of injection
* Bleeding diathesis
* Known allergy to any drugs used

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Effect of caudal nalbuphine on postoperative emergence agitation according to Pediatric Anasthesia emergence delirium (PAED) | Up to 2 hours postoperative
  PAED ( The pediatric anesthesia emergence delirium scale)

SECONDARY OUTCOMES:
Postoperative pain assessment according to Modified Children's Hospital of Eastern Ontario Pain Scale (modified CHEOPS) | For 24 hours postoperative

IPD SHARING:
Plan to Share IPD: Undecided